CLINICAL TRIAL: NCT06297590
Title: A Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3954068 in Patients With Early Symptomatic Alzheimer's Disease
Brief Title: A First-In-Human Study of LY3954068 in Participants With Early Symptomatic Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18795; J4T-MC-OLAA (Other: Eli Lilly and Company); 2024-510604-37-00 (Other: EU Trial Number); U1111-1302-6222 (Other: Universal Trial Number)
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Tau; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Pick Disease of the Brain; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Cognitive Dysfunction | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3954068 (Part A) (Experimental): Single ascending dose of LY3954068 administered intrathecally (IT)
  Interventions: Drug: LY3954068; Drug: Flortaucipir F18
- Placebo (Part A) (Placebo Comparator): Single ascending dose of placebo administered IT
  Interventions: Drug: Placebo; Drug: Flortaucipir F18
- LY3954068 (Part B) (Experimental): Multiple ascending dose of LY3954068 administered IT
  Interventions: Drug: LY3954068; Drug: Flortaucipir F18
- Placebo (Part B) (Placebo Comparator): Multiple ascending dose of placebo administered IT
  Interventions: Drug: Placebo; Drug: Flortaucipir F18

INTERVENTIONS:
Drug: LY3954068 — Administered IT
  Arms: LY3954068 (Part A); LY3954068 (Part B)
Drug: Placebo — Administered IT
  Arms: Placebo (Part A); Placebo (Part B)
Drug: Flortaucipir F18 — Administered intravenously (IV) prior to Positron Emission Tomography (PET) scan

SUMMARY:
The main purpose of this study is to evaluate the safety of LY3954068 in participants with early symptomatic Alzheimer's Disease (AD). The study will also investigate how much LY3954068 gets into the bloodstream and will test the effects of LY3954068 on markers of AD.

The study will be comprised of two parts, A and B. Each enrolled participant in Part A will receive a single dose of LY3954068 or placebo (no active drug) given into the spinal fluid. Each participant in Part B will receive 2 doses of either LY3954068 or placebo administered into the spinal fluid. Participants will have the opportunity to join an optional bridging period to a separate potential study where participants would receive LY3954068.

The study will last up to approximately 45 weeks for Part A, and 100 weeks for Part B, including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) within the range 18 to 40 kilograms per square meter (kg/m²), inclusive, at screening.
* Have gradual and progressive change in memory function for greater than or equal to (≥) 6 months as reported by the participant or informant.
* Have a mini mental state examination (MMSE) score of 18 to 30 at screening.
* Have a clinical dementia rating (CDR) global score of 0.5 to 1.0, with a memory box score ≥ 0.5 at screening.
* Meet flortaucipir F18 positron emission tomography (PET) criteria, as defined in the TAUVID™ FDA label (TAUVID™ prescribing information, 2024), demonstrating evidence of tau pathology.
* Males who agree to follow contraceptive requirements, or women not of childbearing potential (WNOCBP).
* Participants must have up to 2 study partners who are with contact with the participant at least 10 hours per week and one of whom can attend study appointments.

Exclusion Criteria:

* Has current serious or unstable illnesses including cardiovascular, hepatic, renal, gastroenterological, respiratory, endocrinologic, neurologic (other than Alzheimer's Disease), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses in this study; or has a life expectancy of less than (<)24 months.
* Have a sensitivity to flortaucipir F18.
* Have contraindication to magnetic resonance imaging (MRI), including claustrophobia or the presence of contraindicated metal (ferromagnetic) implants/cardiac pacemaker.
* Have a current exposure to an amyloid targeted therapy (ATT). Prior exposure to ATTs greater than 1 year from the last dose may be permitted at the discretion of the investigator and in consultation with the sponsor.
* Have previous exposure to any Investigational Medicinal Product administered intrathecal (IT) or previous exposure to any anti-tau therapy.
* Have a history of clinically significant back pain, back pathology and/or back injury (for example, degenerative disease, spinal deformity or spinal surgery) that may predispose to complications or technical difficulty with lumbar puncture.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of participants with one or more Adverse Event (s) (AEs), Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) considered by the investigator to be related to study drug administration | Baseline up to Week 24 and Week 72 (for optional bridging period participants)
  A summary of AEs, TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the reported adverse events module
Part B: Number of participants with one or more Adverse Event (s) (AEs), Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) considered by the investigator to be related to study drug administration | Baseline up to Week 52
  A summary of AEs, TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the reported adverse events module

SECONDARY OUTCOMES:
Part A: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) | Day 1 up to Week 24
  To evaluate plasma concentration of LY3954068
Part B: PK: Cmax | Day -1 up to Week 52
  To evaluate plasma concentration of LY3954068
Part A: PK: Area Under the Concentration Versus Time Curve (AUC) | Day 1 up to Week 24
  To evaluate plasma concentration of LY3954068
Part B: PK: AUC | Day -1 up to Week 52
  To evaluate plasma concentration of LY3954068
Part A: PK: Cerebrospinal Fluid (CSF) concentration of LY3954068 | Day 3 up to Week 24
  To evaluate CSF concentration of LY3954068
Part B: PK: CSF concentration of LY3954068 | Day 3 up to Week 52
  To evaluate CSF concentration of LY3954068
Part A: Pharmacodynamics (PD): Change from Baseline of CSF tau | Baseline up to Week 24
  To evaluate the effect of LY3954068 on CSF tau
Part B: PD: Change from Baseline of CSF tau | Baseline up to Week 52
  To evaluate the effect of LY3954068 on CSF tau

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (6):
  - K2 Medical Research, LLC, Maitland, Florida
  - Charter Research, LLC, The Villages, Florida
  - CenExel iResearch, LLC (CenExel iRA), Decatur, Georgia
  - Massachusetts General Hospital (MGH), Charlestown, Massachusetts
  - CenExel AMRI, Toms River, New Jersey
  - Duke University, Durham, North Carolina
- The University of Tokyo Hospital, Bunkyō City, Japan
- United Kingdom (3):
  - National Hospital for Neurology and Neurosurgery (UCLH), London
  - Royal Hallamshire Hospital, Sheffield
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A First-In-Human Study of LY3954068 in Participants With Early Symptomatic Alzheimer's Disease — https://trials.lilly.com/en-US/trial/466315